CLINICAL TRIAL: NCT01273987
Title: Neobladder Posterior Wall Suspended With Round Ligament of Uterus After Radical Cystectomy in Female With Bladder Cancer -a Prospective Control Study
Brief Title: Neobladder Posterior Wall Suspended With Round Ligament of Uterus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhiwen Chen (Other)
Responsible Party: Sponsor-Investigator, Zhiwen Chen, Vice director of urological institiute of PLA, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neobladder-01
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Female; Bladder Cancer; Radical Cystectomy; Neobladder; Posterior Wall Suspended With Round Ligament of Uterus
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- neobladder with round lig (Experimental): ileal neobladder suspened with round ligament
  Interventions: Procedure: rONB
- standard neobladder (No Intervention): conventional standard neobladder

INTERVENTIONS:
Procedure: rONB — Neobladder posterior wall suspended with round ligament of uterus after radical cystectomy in female with bladder cancer
  Arms: neobladder with round lig

SUMMARY:
Objective: to evaluate if the Neobladder posterior wall suspended with round ligament of uterus could improve neobladder empty after radical cystectomy in female patients with bladder cancer compared to present standard neobladder

DETAILED DESCRIPTION:
The investigators developed a technical modification which to aim to provide an posterior support to the ideal neobladder and obtain the anatomy recovered neobladder by posterior wall of neobladder suspended with round ligament. In this study the investigators designed the prospective random trial to evaluate whether this technique improves the neobladder empty compared to a current standard neobladder reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were bladder cancer (Stage T1G3, T2-3N0-NxM0), female (age between 40 and 70 years old), no history of urethral trauma or urethral stricture; and a desire to obtain an orthotopic neobladder

Exclusion Criteria:

* The exclusion criteria were male sex, posterior urethral margin confirmed as cancer invasive by pathology; and enteritis. The indications and contraindications for orthotopic reconstruction in this study conformed to the criteria set by the guidelines of the European Association of Urology on bladder cancer

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
postvoiding residual urine (PVP) | 2 years after operation
  number of patients with postvoiding residual urine (PVP) more than 100ml
clean intermittent catheterization(CIC) | 2 years after operation
  number of patients required clean intermittent catheterization(CIC)

SECONDARY OUTCOMES:
rate of complication | through study completion, an average of 2 years
  number of patients with any complication
urodynamic profile | 12 months afer operation
  urodynamic parameter including peak flow rate, functional urethral length ...etc
rate of continence of neobladder | 12 months after operation
  number of patients with continence at daytime and nighttime

CONTACTS AND LOCATIONS:
Overall Officials: ZhiWen Chen, M.D., Study Chair — Urology Institute of PLA, Southwest Hospital, Chongqin, China; HuiXiang Ji, M.D., Principal Investigator — Urology Institute of PLA, Southwest Hospital, Chongqin, China
Locations (1):
- Urology Institute of PLA, Southwest Hospital, Chongqing, China